CLINICAL TRIAL: NCT00491296
Title: Changes in Prostate Specific Antigen Levels During Synergo Therapy-Intravesical Chemotherapy Instillations Combined With Hyperthermia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 0034-07-EMC
Record Dates: First submitted 2007-06-19; First posted 2007-06-26 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2007-06

CONDITIONS: Bladder Cancer
Keywords: S/P Transuretral resection of bladder tumor; Recurrent tumor after BCG Treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Diathermy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SYNERGO
Device: SYNERGO-intravesical chemotherapy instillation combined with hyperthermia

SUMMARY:
PURPOSE: We determined whether Synergo therapy- intravesical chemotherapy instillation combined with hyperthermia instillation is associated with elevated prostate specific antigen (PSA). MATERIALS AND METHODS: We will treat 25 consecutive patients with bladder cancer with a 6-week course of Synergo therapy, followed by cystoscopy at 6 weeks. Blood samples for PSA determination will obtain before each synergo therapy application and at cystoscopy with each patient also serving as a control.

Evaluating changes in PSA level in patients undergoing treatment with Synergo delivered local hyperthermia combined with intravesical instillation of Mitomycin C for adjuvant treatment or pt. with recurrent tu of bladder post TURT with BCGtreatment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent transitional cell carcinoma of urinary bladder post endoscopic resection
* PSA Prior synergo therapy application<10
* Normal rectal examination
* Patients willing to sign informed consent according

Exclusion Criteria:

* History of prostate cancer
* Previous history of TCC stage T2 or higher
* Invasive tu of bladder
* Prior pelvic radiotherapy or systemic chemotherapy
* Active prostatitis
* Active tuberculosis

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Study Completion 2007-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: PEREZ DORON, M.D., Principal Investigator — HAEMEK MEDICAL CENTER, UROLOGY DEPARTMENT; Perez Doron, M.D, Principal Investigator — haemek medical center
Locations (2):
- Israel (2):
  - Haemek MC, Afula
  - Department of urology, Afula